CLINICAL TRIAL: NCT02989779
Title: NK1 Antagonists for Pathological Aggression: A Protocol for Harmful, Impulsive, and Self-/Aggressive Behavior (AHIMSA-1) Trial
Brief Title: Neurokinin (NK) 1 Antagonist for Pathological Aggression for Harmful, Impulsive, and Self-/Aggressive Behaviour
Acronym: AHIMSA-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Gary Chaimowitz, Local Primary Investigator, Head of Forensics, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-1986-GRA
Record Dates: First submitted 2016-11-23; First posted 2016-12-12 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Aggression
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active/Placebo crossover (Experimental): NK1 Antagonist 7 days followed by placebo 7 days.
  Interventions: Drug: NK1 Antagonist; Drug: Placebo Oral Capsule
- Placebo/Active Crossover (Active Comparator): Placebo for 7 days followed by NK1 Antagonist 7 days.
  Interventions: Drug: NK1 Antagonist; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: NK1 Antagonist
Drug: Placebo Oral Capsule

SUMMARY:
Neurokinin (NK) -1 antagonist will be administered to study patients in a double-blind placebo trial. Patients receive assessments including Anger Disorder Scale (ADS) and Modified Overt Aggression Scale (MOAS) and perform computerized study tasks during MRI before the trial begins. Patients receive either one week of the drug or one week of placebo and perform the same tasks and assessments. Then patients receive another week of the alternate pill, followed by another round of tasks during MRI and assessments.

ELIGIBILITY:
Inclusion Criteria:

* are outpatients between 18 and 65 years old inclusive
* meet diagnostic criteria for either Intermittent Explosive Disorder or the adult-modified criteria for Disruptive Mood Dysregulation Disorder (Appendix A)
* have maintained a stable regimen of psychotropic medications (antidepressants, antipsychotics, anticonvulsants, and anxiolytics) for at least 4 weeks prior to study enrolment and throughout the duration of the treatment phase of the study
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
* Have capacity with respect to medical decision-making and consent to participate
* pass the TMS Assessment Safety Survey (TASS) MRI safety questionnaire

Exclusion Criteria:

* have a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or other primary psychotic disorder
* meet criteria for a current manic episode or hypomanic episode
* have a diagnosis of dementia or other neurodegenerative illness affecting the central nervous system
* have a history of substance dependence or abuse within the last 3 months
* are pregnant or currently nursing*

  * *Patients will be tested before and after the study with a urine pregnancy test.
* are taking contraindicated or interacting medications from product monograph of aprepitant
* have an implanted intracranial device or pacemaker
* have a diagnosis of severe hepatic insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Overt Aggression Scale | 1 week

SECONDARY OUTCOMES:
Change in Ball passing task | 1 week
  computer task
Change in Point Subtraction Aggression Task (PSAT) | 1 week
  Computer task
Change in Anger Disorders Scale (ADS) | 1 week
Change in Buss-Perry Aggression Questionniare (BPAQ) | 1 week
Change in State-Trait Anger Expression Inventory | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified information will be shared with University Health Network, Toronto Western Hospital (UHN-TWH) for analysis, as a collaboration site.